CLINICAL TRIAL: NCT02549495
Title: Evaluation of a Community Health Worker Intervention on Adherence to Therapy for Non-Communicable Chronic Disease in Chiapas, Mexico
Brief Title: Impact of Community Health Workers on Adherence to Therapy for Non-Communicable Chronic Disease in Chiapas, Mexico
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Daniel Palazuelos, Associate Physician, Brigham and Women's Hospital
Other Study IDs: 2013P000711
Record Dates: First submitted 2015-04-17; First posted 2015-09-15 (Estimated); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Diabetes or Hypertension: All patients in the seven study communities will receive the community health worker intervention provided by CES, as it is incorporated into the standard of care. However, they will receive the intervention at different points in time depending on which community they lived in, as community health worker programs can only be started at every-three-month intervals

SUMMARY:
This study evaluates the effectiveness of community health workers when added to routine care for patients with diabetes and high blood pressure in rural clinics in Chiapas, Mexico. It does so by recording information on adherence to therapy, blood pressure and hemoglobin A1c while a non-governmental organization working in Mexico trains and introduces a community health worker program.

DETAILED DESCRIPTION:
Compañeros en Salud (CES), an affiliate project of Partners in Health, has been working in the rural Sierra of Chiapas, Mexico since February 2012. CES works in partnership with the local Ministry of Health to rehabilitate and staff existing government primary care clinics. Each community's clinic is staffed by one CES project physician year-round. CES activities span the range of allopathic medicine, but the focus of the project is in the prevention, detection, diagnosis and management of non-communicable diseases (NCDs) such as diabetes and hypertension. CES currently operates in several rural communities with catchment areas of approximately 1,500 - 2,500 people. Routine care for NCDs is based on national guidelines and consists of monthly in-clinic visits by primary care physicians.

Over 9 months in 2014 and again over 6 months in 2016, CES will introduce a community health worker program called "Acompañantes" to its project communities to augment care of patients with NCDs. Acompañantes are lay health workers and members of the community who bridge the gap between project clinics and patients, improving understanding of NCDs, their treatments, and adherence to therapy. The introduction of Acompañantes to communities is planned in a once-every-three-months fashion, the most rapid roll-out logistically feasible for CES. The investigators' project will document their experience over this time, and for one year after introduction of the Acompañantes program to all seven study communities, by documenting adherence to therapy, hemoglobin a1c, and blood pressure at every-three month intervals over this time frame.

ELIGIBILITY:
Inclusion Criteria:

* Formal diagnosis of Type II Diabetes Mellitus, Stage I or II Hypertension or both
* Daily medications required for patient's condition
* Residence and receipt of therapy within the study catchment area
* Age greater than or equal to 18 years.

Exclusion Criteria:

* Known or suspected secondary hypertension
* Known or suspected Type 1 diabetes
* Pregnancy
* Chronic use of glucocorticoids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with Diabetes Mellitus, Type 2, or Hypertension, taking daily therapy, living in one of seven study communities in rural Chiapas, Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2013-03; Primary Completion 2018-04 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Newman, MD, Study Director — Brigham and Women's Hospital; Daniel Palazuelos, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Worster DT, Franke MF, Bazua R, Flores H, Garcia Z, Krupp J, Maza J, Palazuelos L, Rodriguez K, Newman PM, Palazuelos D. Observational stepped-wedge analysis of a community health worker-led intervention for diabetes and hypertension in rural Mexico. BMJ Open. 2020 Mar 8;10(3):e034749. doi: 10.1136/bmjopen-2019-034749. PMID 32152172
- [Result] Newman PM, Franke MF, Arrieta J, Carrasco H, Elliott P, Flores H, Friedman A, Graham S, Martinez L, Palazuelos L, Savage K, Tymeson H, Palazuelos D. Community health workers improve disease control and medication adherence among patients with diabetes and/or hypertension in Chiapas, Mexico: an observational stepped-wedge study. BMJ Glob Health. 2018 Feb 15;3(1):e000566. doi: 10.1136/bmjgh-2017-000566. eCollection 2018. PMID 29527344

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with diabetes, hypertension and respective risk factors were identified via a CES programme of clinic-based and door-to-door case finding.
Pre-assignment Details: Patients were excluded from participation after enrollment but prior to start of study if they were taken off treatment, we not actually on treatment, were enrolled after baseline data collection, moved outside study area, sought care in a different health system, or were found not to have diabetes and/or hypertension.
Groups:
- Patients With Diabetes or Hypertension: All patients in the seven study communities will receive the community health worker intervention provided by CES, as it is incorporated into the standard of care. However, they will receive the intervention at different points in time depending on which community they lived in, as community health worker programs can only be started at every-three-month intervals. Due to the stepped programmatic roll-out, the study mimics a stepped wedge cluster-randomized trial.
Period: Overall Study
Arm/Group | Patients With Diabetes or Hypertension
Started | 168
Completed | 127
Not Completed | 41
Not completed — Death | 2
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 22
Not completed — Lost to Follow-up | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Diabetes or Hypertension
Number analyzed (Participants) | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 107
  >=65 years | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [50 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 149
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 149
Has a radio [Count of Participants; unit: Participants] | 93
Has a car/motorcycle [Count of Participants; unit: Participants] | 43
Type of remuneration [Count of Participants; unit: Participants]
  Salary | 8
  Day labour | 58
  None | 83
Diabetes diagnosis [Count of Participants; unit: Participants] | 70
Hypertension diagnosis [Count of Participants; unit: Participants] | 110
Systolic Blood Pressure [Median (Inter-Quartile Range); unit: mm Hg] | 135 [126 to 151]
HbA1c [Median (Inter-Quartile Range); unit: percent of glycosylated hemoglobin] | 9.3 [7.2 to 11.7]

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c
Description: Change in percent glycated hemoglobin as measured by PTS diagnostics point-of-care assay
Time Frame: Baseline, 23 months
Measure: Median (95% Confidence Interval); unit: percentage of glycated hemoglobin
Groups:
- Patients With Diabetes: Patients with diabetes included in the study
Arm/Group | Patients With Diabetes
Number analyzed (Participants) | 73
percentage of glycated hemoglobin | -0.35 [-0.90 to 0.2]

2. Primary Outcome: Change in Systolic Blood Pressure
Description: Change in Systolic blood pressure as measured by Omron HEM 7080IT electronic blood pressure monitor
Time Frame: Baseline, 23 months
Measure: Median (95% Confidence Interval); unit: mmHg
Groups:
- Patients With Hypertension: Patients with hypertension included in the study
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 117
mmHg | -4.7 [-8.9 to -0.6]

3. Secondary Outcome: Change in Adherence to Daily Medications
Description: Change in self-reported medication adherence as measured by 5-day recall, 30-day recall and response to Likert-style questions
Time Frame: One year after all communities receive intervention
Population: Data were not collected for this measure and the outcome cannot be reported
Groups:
- Patients With Diabetes or Hypertension: All patients with diabetes and/or hypertension
Arm/Group | Patients With Diabetes or Hypertension
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure as measured by Omron HEM 7080IT electronic blood pressure
Time Frame: Baseline, 23 months
Measure: Median (95% Confidence Interval); unit: mmHg
Arm/Group | Patients With Hypertension
Number analyzed (Participants) | 117
mmHg | -2.2 [-4.5 to 0.1]

5. Secondary Outcome: Disease Control
Description: Diabetes and/or hypertension control. Disease control among patients with hypertension was defined according to Mexican national guidelines: blood pressure <140/90 mm Hg for patients with hypertension and no diabetes; blood pressure <130/80 mm Hg for patients with hypertension and diabetes and blood pressure < 150/90 mm Hg for patients over the age of 80. Disease control for patients with diabetes defined as glycated hemoglobin (HbA1c) < 7% per national guidelines.
Time Frame: One year after all communities receive intervention
Population: Data were not collected and the outcome cannot be reported
Arm/Group | Patients With Diabetes or Hypertension
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 2 years
Description: Study staff regularly monitored participants and kept an adverse event log that was reported to the IRB. Clinical events monitored include death, myocardial infarction, and stroke.
Groups:
- Standard of Care: Patients with hypertension and/or diabetes across seven study communities prior to CHW intervention.
- CHW Intervention: Patients with hypertension and/or diabetes across seven study communities following CHW intervention.
Arm/Group | Standard of Care | CHW Intervention
All-Cause Mortality (participants affected / at risk) | 1/149 | 1/149
Serious Adverse Events (participants affected / at risk) | 0/149 | 1/149
Other Adverse Events (participants affected / at risk) | 0/149 | 0/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=149) | CHW Intervention (N=149)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1) — Coronary artery disease would not be expected to result from standard of care or the intervention
Stroke (Nervous system disorders) | 0 (0) | 0 (0) — Stroke would not be expected to result from standard of care or the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/95/NCT02549495/Prot_SAP_000.pdf